CLINICAL TRIAL: NCT04716907
Title: Thymic Function in Patients With COVID-19
Acronym: COVITHYM
Status: Completed | Type: Observational
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/06
Record Dates: First submitted 2021-01-16; First posted 2021-01-20 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Covid19
Keywords: Covid19; Thymic function; Genetic polymorphism
MeSH Terms: conditions — COVID-19 | interventions — Polymorphism, Single Nucleotide; Blood Specimen Collection; Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case : COVID-19 positive patients: patients hospitalized for COVID-19 infection
  Interventions: Genetic: Single-Nucleotide Polymorphisms (SNP) within the TCRA/D region; Biological: Blood sample; Diagnostic Test: CT Scan; Biological: Bronchial fibroscopy
- Control : COVID-19 negative patients: patients hospitalized for other reasons
  Interventions: Biological: Blood sample; Diagnostic Test: CT Scan

INTERVENTIONS:
Genetic: Single-Nucleotide Polymorphisms (SNP) within the TCRA/D region — DNA extraction from blood samples, PCR and Sequencing
  Groups: Case : COVID-19 positive patients
Biological: Blood sample — Dosage of sj/βTREC ratio, lymphocytes, cytokines and chemokines.
Diagnostic Test: CT Scan — Thymus and lung imaging
Biological: Bronchial fibroscopy — Bronchoalveolar lavage in mechanically ventilated patients for dosage of recent thymic emigrants in lungs
  Groups: Case : COVID-19 positive patients

SUMMARY:
The main clinical manifestation associated with SARS-CoV-2 infection is an influenza-like illness that follows the infection of the respiratory tract. In a few percent of infected people, inflammation of the lungs leads to severe pneumonia that requires hospitalization, in intensive care units for the more severe cases. Despite intensive care, a fatal outcome occurs in 6% and 12% of women and men over 80 years of age hospitalized for severe COVID, respectively.

Factors associated with a higher risk of death in patients with SARS-CoV-2 include age and low circulating lymphocyte counts. Significant lymphopenia is indeed frequently observed in patients with severe COVID-19 and both phenotypic and functional changes in antiviral T cells have been correlated with the severity of COVID-19.

The thymus, the organ that produces T lymphocytes, undergoes progressive physiological involution with age. However, in the elderly, rare cases of thymic hyperplasia are reported in autoimmune diseases or cancers, or are observed in response to deep lymphopenia, whether or not associated with sepsis.

This cohort of patients treated for a SARS-CoV-2 infection could allow to better understand the role of the thymus in this pathology.

ELIGIBILITY:
Inclusion Criteria:

Cases :

* Patients with confirmed COVID-19 infection
* Hospitalized for COVID-19 infection
* Having signed a written informed consent form
* Affiliation to the social security system

Controls :

* Non-COVID-19 patients
* Hospitalized for other reasons
* Age and sex-matched controls
* Having signed a written informed consent form,
* Affiliation to the social security system

Exclusion Criteria:

* Autoimmune disease
* HIV, Hepatitis B or Hepatitis C
* Pregnant or breastfeeding women
* A mental or linguistic inability to understand the study
* Patient under protection of the adults (guardianship, curators or safeguard of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 50 cases and 50 control subjects
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2022-04-02 (Actual); Study Completion 2022-04-02 (Actual)

PRIMARY OUTCOMES:
Genetic Predisposition to severe forms of COVID-19 | through study completion, average 1 year
  Test of association between single-nucleotide polymorphisms (SNP) within the TCRA/D region known to influence the level of thymopoiesis (Clave et al., Sci Transl Med., 2018) and CT scan classification of COVID-associated pneumopathy (0=Absent or minor pulmonary parenchymal changes ; 1=Limited ground-glass opacities ; 2=Bilateral ground-glass opacities < 50% of pulmonary parenchyma ; 3=Idem 2, with superimposed inter/intra lobular septal thickening, i.e. 'crazy paving' ; 4=Bilateral ground-glass opacities > 50% of pulmonary parenchyma ; 5=Idem 4, with superimposed 'crazy paving' ; 6=Idem 5, with pulmonary fibrosis).

SECONDARY OUTCOMES:
Genetic Predisposition to thymic enlargement observed during COVID-19 infection | through study completion, average 1 year
  Test of association between single-nucleotide polymorphisms (SNP) within the TCRA/D region known to influence the level of thymopoiesis (Clave et al., Sci Transl Med., 2018) and CT scan classification of thymus aspects (0=Fatty thymus atrophy (the most common in middle aged adults) ; A=Homogeneous non-fatty thymus (common in young adults) or Fat in the thymus area associated with micronodules or Moderate infiltration of the thymus area ; B=Hyperplasia, marked infiltration, micronodules or Hyperplasia with well-defined contours or Nodular hyperplasia without a tumour mass or Pseudo-tumoral mass with well-defined contours).
Genetic Predisposition to enhanced thymic function during COVID-19 infection | through study completion, average 1 year
  Test of association between single-nucleotide polymorphisms (SNP) within the TCRA/D region known to influence the level of thymopoiesis (Clave et al., Sci Transl Med., 2018) and sj/βTREC ratio.
Genetic Predisposition to severity of COVID-19 pathology | through study completion, average 1 year
  Test of association between single-nucleotide polymorphisms (SNP) within the TCRA/D region known to influence the level of thymopoiesis (Clave et al., Sci Transl Med., 2018) and ICU length of stay.
Basal thymic function in COVID patients | through study completion, average 1 year
  Analysis of sj/βTREC ratio during infection and away from infection (> 6 months).
Thymic function in COVID patients | through study completion, average 1 year
  Analysis of sj/βTREC ratio in COVID positive patients and in COVID negative patients
Immune response in COVID patients | through study completion, average 1 year
  Analysis of lymphocytes in COVID positive patients and in COVID negative patients
Immune response in lungs of COVID patients | through study completion, average 1 year
  Analysis of recent thymic emigrants in the bronchoalveolar fluid of COVID positive patients
Inflammatory response in COVID patients | through study completion, average 1 year
  Analysis of serum concentrations of cytokines and chemokines in pg/ml (composite : IFNα, IFNβ, IL-17A, IL17F, IL21, IL22, IL23, IL27, IL29, TSLP, GM-CSF, IL10, IL12p70, IL1β, IL4, IL6, TNFα, VEGF, IL15, IL17E, IL33, IL8, MDC, Mip1α, Mip1β, Mip3α, SDF1), in COVID positive patients and in COVID negative patients

CONTACTS AND LOCATIONS:
Locations (1):
- CMC Ambroise Paré, Neuilly-sur-Seine, France

IPD SHARING:
Plan to Share IPD: No